CLINICAL TRIAL: NCT06337045
Title: Atrial Fibrillation and Municipality-based Prevention and Rehabilitation - a Feasibility Study
Brief Title: Atrial Fibrillation, Prevention and Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Department of Cardiology, Odense University Hospital, Odense, Denmark. (Unknown); Health Center, Municipality of Svendborg, Svendborg, Denmark. (Unknown); Department of Internal Medicine & Emergency Department, Svendborg Hospital, Odense University Hospital, Svendborg, Denmark. (Unknown); The Danish Heart Association, Funen, and local committee in Svendborg, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AF-rehab
Record Dates: First submitted 2024-02-27; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Prevention; Rehabilitation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Eligible participants were diagnosed with AF at the hospital and had symptomatic AF rated by the modified European Heart Rhythm Association (mEHRA) score ≥2B. If the patient was eligible based on the mEHRA-score, at least one of the following risk factors had to be present: hypertension, diabetes, obesity, smoking, excessive alcohol consumption, physical inactivity, sleep apnoea, anxiety, depression, or mental vulnerability.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complex prevention and rehabilitation intervention (single arm) (Experimental): It was a single-arm study.
  Interventions: Behavioral: Complex prevention and rehabilitation intervention

INTERVENTIONS:
Behavioral: Complex prevention and rehabilitation intervention — The complex intervention started and ended with individual consultations with health professionals and furthermore included physical exercise, smoking cessation, alcohol treatment, dietary interventions, AF specific patient education, MediYoga, and/or psychosocial support.

SUMMARY:
Evidence shows that people with atrial fibrillation (AF) can benefit from prevention and rehabilitation interventions related to quality of life, lowered anxiety, etc. In this study, a complex prevention and rehabilitation intervention for people with AF was carried out in a Health Center at a Danish municipality in cooperation with the cardiology department at Svendborg Hospital. The study was designed as a feasibility study, with data gathered systematically including focus group interviews and quantitative patient reported outcomes. People with AF were included at the hospital. Eligible participants were offered intervention in the Health Center. Interventions, in accordance with present international guidelines, consisted of physical exercise, patient education, psychosocial support and consultations with health professionals as well as risk factor management. Also, medicinal yoga (MediYoga) were chosen to be part of the intervention due to promising research results within AF. All interventions were optional and based on needs assessment and preferences.

The primary objective was to investigate the feasibility of delivering a complex prevention and rehabilitation intervention for people with AF in a municipal Health Center.

There were the following four secondary objectives:

1. To explore the participant's experiences of participating in the municipality-based complex prevention and rehabilitation intervention.
2. To explore the participant's needs and preferences of the interventions.
3. To explore changes in HRQoL, anxiety and depression.
4. To explore the feasibility of collecting patient reported outcome measures as part of the intervention.

The hypothesis was that the complex prevention and rehabilitation intervention was feasible in a municipality-based set-up, and was well received by people with AF and may contribute to better outcomes in terms of HRQoL, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* the modified European Heart Rhythm Association (mEHRA) score ≥2B.

And at least one of the following risk factors:

* Hypertension (treatment with >1 drug, diagnosis verified by home-blood pressure measurement, 24-hour ambulatory blood pressure measurement, or consultation blood pressure measurement >160/90mmHg).
* Diabetes mellitus (HbA1c > 58mmol/mol unless higher values are accepted due to other aspects).
* Obesity (Body Mass Index > 30).
* Smoking (active smoker).
* Alcohol consumption (> 7 units per week for women and > 14 units per week for men (according to the Danish Health Authority guidelines from 2019), or motivation for reduction).
* Physical inactivity (less than the recommended 30 minutes per day).
* Known sleep apnea or STOP-bang Sleep Apnea Questionnaire score >3).
* Symptoms of anxiety or depression evaluated by the Hospital Anxiety and Depression Scale (HADS) > 7.
* Mental vulnerability defined as self-evaluated burdened life with high perceived stress, small social network, and/or low educational level.

Exclusion Criteria:

* ongoing treatment adjustments due to heart failure.
* ongoing cardiac rehabilitation.
* dementia, mental illness, language barrier or comorbidity that made it impossible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
HeartQoL | HeartQoL was collected at three time points: T0 (baseline), T1 (end of intervention, an average of 4 months) and T2 (follow-up 2-months later). The intervention phase (T0 to T1) was individual based on needs assessment.
  HeartQoL measures Health-related Quality of Life (HRQoL). HeartQoL contains three scales, a global overall scale and a physical- and emotional sub-scale. It has a 14-item self-assessment scale enabling the respondents to recall how much their heart problem have bothered them during the past four weeks on a 4-point Likert scale from 0-3, where higher score represents better HRQoL. The global score reflects all items and is calculated by dividing the sum of the scored items by the number of scored items. The same principle goes for the physical- and emotional subscales, which respectively holds 10 items and 4 items.
The hospital anxiety and depression scale (HADS) | HADS was collected at three time points: T0 (baseline), T1 (end of intervention, an average of 4 months) and T2 (follow-up 2-months later). The intervention phase (T0 to T1) was individual based on needs assessment.
  HADS measures symptoms of anxiety and depression. HADS is a 14-item self-assessment scale, 7 items for each domain. All items are rated on a 4-point Likert scale, where 0 reflects the positive extreme and 3 reflects the negative extreme of the scale. For each domain a score ranging from 0 to 21 can be obtained, and categorized as "normal" (0-7 points), "possible presence of a disorder" (8-10 points), and "probable presence of a disorder" (11-21 points).
Experience of participating, experiences needs and preferences of interventions | Focus group interviews was conducted at T1 (end of intervention, an average of 4 months).
  These data was obtained from focus group interviews.
Feasibility of collecting patient reported outcomes (PROMs). The PROMs was the HeartQoL and the hospital anxiety and depression scale. | Field notes was collected at T2 (follow-up 2 months later).
  These data was obtained from collecting field notes from Health Professionals conducting the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Cardiology, Odense University Hospital, Odense, Region Syddanmark
  - Health Center, Municipality Svendborg, Svendborg, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elnegaard CM, Pedersen MK, Zwisler AO, Borregaard B, Eilso JF, Sommer T, Tveskov C, Hendriks JM, Brandes A, Risom SS. Atrial fibrillation and primary care prevention and rehabilitation - a feasibility study. Pilot Feasibility Stud. 2025 Nov 26;11(1):150. doi: 10.1186/s40814-025-01724-3. PMID 41299666